CLINICAL TRIAL: NCT05485818
Title: Phase IIa Clinical Study of Efficacy and Safety of Injectable Recombinant Human Thymosin Beta 4 in Patients With Acute Myocardial Infarction
Brief Title: Safety and Efficacy Study of Thymosin Beta 4 in Patients With Acute Myocardial Infarction.Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL005-AMI-IIa
Record Dates: First submitted 2020-09-07; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Acute Myocardial Infarction
Keywords: AMI
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): Patients in this treatment group will receive NL005 for 0.25 ug/kg respective.Continuous administration for 7 days.
  Interventions: Drug: Low Dose
- Middle Dose (Experimental): Patients in this treatment group will receive NL005 for 0.5 ug/kg respective.Continuous administration for 7 days.
  Interventions: Drug: Middle Dose
- High Dose (Experimental): Patients in this treatment group will receive NL005 for 2.0 ug/kg respective.Continuous administration for 7 days.
  Interventions: Drug: High Dose
- Placebo (Placebo Comparator): Patients in this treatment group will receive placebo respective. Continuous administration for 7 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Low Dose — 12±4 hours after PCI: 0.25 ug/kg Recombinant Human Thymosin β4 （intravenous injection），Day2-Day7 after PCI：0.25 ug/kg Recombinant Human Thymosin β4 （intravenous injection）
  Other Names: NL005（ Low Dose）
  Arms: Low Dose
Drug: Middle Dose — 12±4 hours after PCI: 0.5 ug/kg Recombinant Human Thymosin β4 （intravenous injection），Day2-Day7 after PCI：0.5 ug/kg Recombinant Human Thymosin β4 （intravenous injection）
  Other Names: NL005（ Middle Dose）
  Arms: Middle Dose
Drug: High Dose — 12±4 hours after PCI: 2.0 ug/kg Recombinant Human Thymosin β4 （intravenous injection），Day2-Day7 after PCI：2.0 ug/kg Recombinant Human Thymosin β4 （intravenous injection）
  Other Names: NL005（High Dose）
  Arms: High Dose
Other: Placebo — 15 subjects will be randomly assigned to the placebo for 7 days
  Arms: Placebo

SUMMARY:
A multicenter randomized double-blind placebo parallel control design was used in this study.60 subjects eligible for inclusion will be randomly assigned to either a low-dose (0.25ug/kg) medium-dose (0.5ug/kg) high-dose (2.0ug/kg) experimental drug group or a control group (placebo) at a ratio of 1:1:1:1.After randomization, subjects received the experimental drug or placebo once a day, intravenously, on day 2 to 7, 12 hours and 4 hours after PCI.Ninety days after PCI were observed.

DETAILED DESCRIPTION:
Subjects underwent cardiovascular magnetic resonance imaging (CMR) on the 90th day after PCI, which was used to evaluate the myocardial salvage index myocardial infarction area, microvascular occlusion area, left ventricular ejection fraction (LVEF), left ventricular end-systolic volume (LVESV), and left ventricular end-diastolic volume (LVEDV).Echocardiography was performed on the 5th and the 90th day after PCI to evaluate the left indoor diameter (LV) and left atrial diameter (LA) of LVEF.

Physical examination routine blood coagulation function was performed on the 30th and 90th day after PCI in the screening period (pre-screening results were acceptable);Electrocardiogram (ECG) was performed on the 30th and the 90th day after PCI on the 2nd day after the first administration;During the screening period (results before screening are acceptable), vital signs should be measured from day 1 to day 7 after PCI (during each dose, vital signs should be measured twice on day 7, including before and after administration), on day 30 and day 90;Blood biochemical examinations were performed from day 2 to day 4, day 7, day 30, and day 90 after PCI before the first administration;Creatine kinase isoenzyme (CK-MB) hypersensitive troponin I(HS-CTNI) or troponin I(cTnI) and amino-terminal B-type natriuretic peptide precursor (NT-probNP) or B-type natriuretic peptide (BNP) were detected on day 2, day 3, day 4 and day 7 after PCI before the first administration.Tumor markers were detected and immunogenicity blood samples were collected 30 days after PCI before the first administration.Routine urinalysis was performed 90 days after PCI before the first administration;Adverse drug events and cardiovascular events were continuously recorded during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or its legal representative will voluntarily participate in the study and sign the informed consent;
2. Age 18 and 75, regardless of gender;
3. STEMI patients with left anterior descending branch single-artery middle occlusion (TIMI grading 0~1, see Appendix 1 for TIMI grading) and receiving PCI;
4. No obvious collateral of coronary artery (Rentrop grade 0~1,Rentrop grade see Appendix 2);
5. Chest pain occurred for 6 hours and 12 hours before PCI;
6. TIMI grade 3 after PCI;
7. All subjects (male and female) must agree to use appropriate contraceptive methods (hormonal or barrier contraceptive methods, abstinence) during the study period and up to 6 months after the last administration, and women of childbearing age must test negative for pregnancy before administration.

Exclusion Criteria:

1. Patients who have a history of myocardial infarction or have received coronary artery acute thrombolytic interventional therapy with bypass surgery;
2. patients who received thrombolytic therapy after onset;
3. patients who were clearly diagnosed as acute heart failure (Killip grade II,Killip classification in annex 3);
4. Severe arrhythmia that cannot be corrected;
5. Aortic dissection or suspected presence;
6. Severe liver and kidney dysfunction or severe depletion, etc;
7. major surgical history or hemorrhagic stroke in half a year;
8. Has or has a history of malignancy;
9. Systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg in patients with hypertension after active antihypertensive treatment;
10. Clinically, he had a significant history of allergy, especially to mannitol, drugs, protein preparations and biological products;
11. Screening of patients who participated in other clinical studies within the first 3 months;
12. Failure to perform CMR test: such as claustrophobia, renal failure (eGFR < 30ml/min);
13. Other conditions not considered suitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Change of myocardial infarction area on Day 5 and day 90 after PCI | Day 5、Day 90
  Change of myocardial infarction area on Day 5 and day 90 after PCI. Myocardial infarction area day 5 and day 90 after PCI，and the change on day 90 compared to day 5. Myocardial infarction size was evaluated by late gadolinium enhanced cardiac magnetic resonance (LGE-CMR) imaging.

SECONDARY OUTCOMES:
Change of myocardial salvage index on Day 5 and day 90 after PCI | Day 5、Day 90
  Myocardial salvage index day 5 and day 90 after PCI，and the change on day 90 compared to day 5. Myocardial salvage index (%) defifined as: (area at risk-infarct size)/ area at risk*100% measured by CMR. Higher scores mean a better outcome.
Change of microvascular obstruction area on Day 5 and day 90 after PCI | Day 5、Day 90
  Area of microvascular obstruction day 5 and day 90 after PCI，and the change on day 90 compared to day 5. Microvascular obstruction is one of the risk factors affecting the prognosis of AMI patients. The occurrence of MVO is related to the release of cytotoxic factors caused by distal microvascular embolization and reperfusion injury. Studies have shown a significantly increased risk of heart failure, adverse cardiovascular events, and death. late gadolinium enhancement (LGE) was performed to identify areas of microvascular obstruction (MVO), the typical MVO is the low signal area in the high signal area of infarction.
Change of LA on Day 5 and day 90 after PCI | Day 5、Day 90
  Change of left atrium (LA) on Day 5 and day 90 after PCI, The data of LA after PCI were measured by CMR at Day 5 and day 90, and calculate changes in data day 90 and day 5.
Changeof LV on Day 5 and day 90 after PCI | Day 5、Day 90
  Change of left ventricle (LV) on Day 5 and day 90 after PCI, Day 5 and day 90 LV after PCIwere measured by CMR at Day 5 and day 90, and calculate changes in data day 90 and day 5.
Change of LVEF on Day 5 and day 90 after PCI | Day 5、Day 90
  Change of Left Ventricular Ejection Fractions (LVEF) on Day 5 and day 90 after PCI, Day 5 and day 90 LVEF after PCIwere measured by CMR at Day 5 and day 90, and calculate changes in data day 90 and day 5.
Change of LVESV on Day 5 and day 90 after PCI | Day 5、Day 90
  Change of Left Ventricular end-systolic volume (LVESV) on Day 5 and day 90 after PCI, Day 5 and day 90 LVESV after PCI were measured by CMR at Day 5 and day 90, and calculate changes in data day 90 and day 5.
Change of LVEDV on Day 5 and day 90 after PCI | Day 5、Day 90
  Change of Left Ventricular end-diastolic volume (LVEDV) on Day 5 and day 90 after PCI, Day 5 and day 90 LVEDV after PCI were measured by CMR at Day 5 and day 90, and calculate changes in data day 90 and day 5.
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0 | Day0、Day1、Day2、Day3、Day4、Day5、Day6、Day7、Day30、Day90
  Number of participants with adverse events (AE), treatment-related adverse events, abnormal vital signs, abnormal physical examination findings, abnormal laboratory test results, abnormal electrocardiograms
Incidence of anti-drug antibody (ADA) | Day 0、Day 30
  Blood samples were collected before administration and 30 days after PCI to evaluate the immunogenicity of NL005

CONTACTS AND LOCATIONS:
Overall Officials: KeFei Dou, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Limana F, Capogrossi MC, Germani A. The epicardium in cardiac repair: from the stem cell view. Pharmacol Ther. 2011 Jan;129(1):82-96. doi: 10.1016/j.pharmthera.2010.09.002. Epub 2010 Oct 19. PMID 20937304
- [Background] Wrigley BJ, Lip GY, Shantsila E. The role of monocytes and inflammation in the pathophysiology of heart failure. Eur J Heart Fail. 2011 Nov;13(11):1161-71. doi: 10.1093/eurjhf/hfr122. Epub 2011 Sep 27. PMID 21952932
- [Background] Gutierrez SH, Kuri MR, del Castillo ER. Cardiac role of the transcription factor NF-kappaB. Cardiovasc Hematol Disord Drug Targets. 2008 Jun;8(2):153-60. doi: 10.2174/187152908784533702. PMID 18537603
- [Background] Gordon JW, Shaw JA, Kirshenbaum LA. Multiple facets of NF-kappaB in the heart: to be or not to NF-kappaB. Circ Res. 2011 Apr 29;108(9):1122-32. doi: 10.1161/CIRCRESAHA.110.226928. PMID 21527742
- [Background] Srivastava D, Ieda M, Fu J, Qian L. Cardiac repair with thymosin beta4 and cardiac reprogramming factors. Ann N Y Acad Sci. 2012 Oct;1270:66-72. doi: 10.1111/j.1749-6632.2012.06696.x. PMID 23050819
- [Result] Dube KN, Bollini S, Smart N, Riley PR. Thymosin beta4 protein therapy for cardiac repair. Curr Pharm Des. 2012;18(6):799-806. doi: 10.2174/138161212799277699. PMID 22236126
- See also: Related info — http://www.northland-bio.com/